CLINICAL TRIAL: NCT03585322
Title: A Phase I Study of the Safety, Pharmacokinetic and Pharmacodynamic Properties of APG-1387 in Patients With Chronic Hepatitis B.
Brief Title: APG-1387 Study of Safety, Tolerability ,PK/PD in Patients With Chronic Hepatitis B
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ascentage Pharma Group Inc. (Industry)
Collaborators: HealthQuest Pharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APG-1387-CN-HBV-001
Record Dates: First submitted 2018-06-26; First posted 2018-07-13 (Actual); Last update posted 2021-11-08 (Actual); Status verified 2021-11

CONDITIONS: Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — APG-1387; Injections

STUDY DESIGN:
Intervention Model Description: dose escalation study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- APG-1387 for Injection (Experimental): APG-1387 will be explored sequentially using a escalation scheme at the dose escalation phase.
  Interventions: Drug: APG-1387 for Injection

INTERVENTIONS:
Drug: APG-1387 for Injection — Multiple dose cohorts, 30 minute IV infusion, once weekly for 4 weeks .

SUMMARY:
This study is a Multiple Ascending Dose study to Explore the Tolerability, Safety and Pharmacokinetics/Pharmacodynamics of APG-1387 in Chronic Hepatitis B Patients.

DETAILED DESCRIPTION:
APG-1387 is a potent, bivalent small-molecule IAP antagonist. This study is multi-center, single-agent, open-label, Phase I dose-escalation study of APG-1387.

This study has a 4-dose-schedule which is escalated one by one after confirming safety in the previous lower dose schedule. A total of 60 subjects with Chronic Hepatitis B will be participated in the study. APG-1387 will be administrated via intravenous infusion, once a week for consecutive 4 weeks as one cycle.The start dose is 7mg. 3 patients' cohorts will be evaluated, the dose of APG-1387 will be increased in subsequent cohorts, to 12mg, 20 mg, 30 mg, 45 mg accordingly. 3 patients in 7mg,12mg cohorts and 6 patients in 20mg, 30mg and 45mg cohorts will be recruited. If there is any one of the following event is observed within 28 days of the first dose of APG-1387, the recruitment will be hold and a discussion on MTD dose level will happened.1 ≥1/2 patients experience ≥Grade 2 toxicities[CTCAE 4.0.3] related or possibly related with APG-1387 and with clinical manifestation. 2 ≥1/3 patients experience ≥Grade 3 toxicities[CTCAE 4.0.3] related or possibly related with APG-1387.3 any SAE related or possibly related with APG-1387. Expansion study will be designed to explore primary efficacy and safety after the dose escalation study. The expansion number and dosage will be decided according to the results of each cohort.(no more than 36 patients).

ELIGIBILITY:
Inclusion Criteria

1. Age ≥18 and ≤ 65 years old.
2. Confirmed diagnosis of chronic hepatitis B, HBsAg positive≥6 months.
3. HBV DNA≥2×103 IU/mL for HBeAg negative patients, HBV DNA≥1×104IU/mL for HBeAg positive patients in screening phase.
4. ALT≥ ULN and <10 ×ULN in screening phase (exclude non-HBV related ALT elevation such as drug or alcohol et al).
5. BMI 18~26.
6. Patients should not use antivirus treatment such as NAs and IFN within 6 months before screening.
7. Adequate hematologic function.
8. QTc interval ≤ 450 ms in males, and ≤ 470 ms in females.
9. Adequate renal and liver function.
10. Negative serum pregnancy test (for women of childbearing potential) documented within the 24-hour prior to the first dose of investigational product. Willing to use contraception by a method that is deemed effective by the investigator by Subject and their partners throughout the treatment period and for at least three months following the last dose of study drug.
11. Ability to understand and willing to sign a written informed consent form, the consent form must be signed by the patient prior to any study-specific procedures.

Exclusion Criteria

1. Clinical confirmed HCC or suspected HCC or AFP>50μg/L.
2. A history of decompensated liver function (such as Child-Pugh B or C or history of ascites, digestive tract bleeding, hepatic encephalopathy or spontaneous bacterial peritonitis et al.).
3. Advanced fibrosis/cirrhosis, defined as a fiber screening scan≥12.4kPa during screening phase or liver biopsy at any time found Metavir score F3, F4 fibrosis.
4. Patients with other liver diseases except hepatitis B, including chronic alcoholic hepatitis, drug-induced liver injury, autoimmune liver disease, hereditary liver disease and other causes of active hepatitis.
5. Patients with malignant tumours (excluding basal cell and in situ cervical cancer that have been cured without recurrence) or lymphatic proliferative diseases.
6. Have a clear history of neurological or psychiatric disorders, such as epilepsy, dementia, poor compliance.
7. Chronic kidney disease, renal insufficiency.
8. Poor control of other important primary diseases of the viscera, such as clear history of nervous system, cardiovascular system, urinary system, digestive system, respiratory system, Metabolism and skeletal muscle system (such as poor control diabetes, hypertension and etc.), which the investigator considers not suitable for the study.
9. Females who are pregnant or nursing.
10. History of alcoholism (average daily ethanol intake of 30 grams (male) or ≥ 20 grams (female) for 1 years), drug abuse history or drug abuse screening results positive.
11. Severe infection, trauma or a major surgical operation within 4 weeks prior to screening.
12. Use of immunomodulators (eg, corticosteroids) or biologics (eg, monoclonal antibody, IFN) within 3 months prior to screening, or will use immunomodulators (eg, corticosteroids) or biologics (eg, monoclonal antibody, IFN) during the study.
13. Treatment with an investigational agent or device within three months prior to screening.
14. Anti-HDV total antibody/IgM antibody positive, HCV antibody positive and HCV-RNA positive, anti-HIV antibody positive, or treponema pallidum antibody positive.
15. Known or suspected Wilson's Disease, or other disease that may affect copper accumulates or regulates.
16. Prior treatment with IAP inhibitors.
17. Any other condition or circumstance of that would, in the opinion of the investigator, make the patient unsuitable for participation in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2018-07-04 (Actual); Primary Completion 2021-10-15 (Actual); Study Completion 2021-10-15 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | 28 days
  Patients with APG-1387 treatment related adverse events (AE), serious adverse events (SAE) will be assessed according NCI CTCAE Version 4.0.3

SECONDARY OUTCOMES:
Pharmacokinetic evaluation | 28 days
  Maximum plasma concentration (Cmax) will be assessed in the patients treated with APG-1387.
Pharmacokinetic evaluation | 28 days
  Area under the plasma concentration versus time curve (AUC) will be assessed in the patients treated with APG-1387 .
Change in serum HBV DNA from baseline at Day 1, Day 8, Day15, Day 22, Day28，Day56，Day84 and Day 112. | Day 1, Day 8, Day15, Day 22, Day28，Day56，Day84，and Day 112
  treatment effects of APG-1387 on Chronic Hepatitis B
Change in serum HBsAg from baseline at Day 1, Day 8, Day15, Day 22, Day28，Day56，Day84 and Day 112. | Day 1, Day 8, Day15, Day 22, Day28，Day56，Day84，and Day 112
  treatment effects of APG-1387 on Chronic Hepatitis B
Change in serum HBeAg from baseline at Day 1, Day 8, Day15, Day 22, Day28，Day56，Day84 and Day 112. | Day 1, Day 8, Day15, Day 22, Day28，Day56，Day84，and Day 112
  treatment effects of APG-1387 on Chronic Hepatitis B
Change in serum HBsAb from baseline at Day 1, Day 8, Day15, Day 22, Day28，Day56，Day84 and Day 112. | Day 1, Day 8, Day15, Day 22, Day28，Day56，Day84，and Day 112
  treatment effects of APG-1387 on Chronic Hepatitis B
Change in serum HBeAb from baseline at Day 1, Day 8, Day15, Day 22, Day28，Day56，Day84 and Day 112. | Day 1, Day 8, Day15, Day 22, Day28，Day56，Day84，and Day 112
  treatment effects of APG-1387 on Chronic Hepatitis B
Change in serum HBcAb from baseline at Day 1, Day 8, Day15, Day 22, Day28，Day56，Day84 and Day 112. | Day 1, Day 8, Day15, Day 22, Day28，Day56，Day84，and Day 112
  treatment effects of APG-1387 on Chronic Hepatitis B

CONTACTS AND LOCATIONS:
Overall Officials: Yifan Zhai, M.D., Ph.D., Study Director — Ascentage Pharma Group Inc.
Locations (2):
- China (2):
  - Nanfang Hospital of Southern Medical University, Guangzhou, Guangdong
  - Guangzhou Eighth People's Hospital, Guangzhou, Guangdong

IPD SHARING:
Plan to Share IPD: No